CLINICAL TRIAL: NCT04225702
Title: Effect Of Long-term Aspirin Preoperative on Postoperative Cognitive Dysfunction In Elderly Patients Undergoing Knee Arthroplasty
Brief Title: Effect Of Aspirin Preoperative on Postoperative Cognitive Dysfunction In Elderly Patients Undergoing Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Jin Dong Liu, Chief physician and Associate Professor, Xuzhou Medical University
Other Study IDs: XYFY2019-KL05
Record Dates: First submitted 2019-10-10; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Elective Surgery; Postoperative Cognitive Dysfunction; Knee Arthroplasty
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Aspirin: The elderly patients who using Aspirin at least three months before operation were in the Group Aspirin
- Group Control: The elderly patients who not using Aspirin before operation were in the Group Control

SUMMARY:
Studies have shown that the lifetime risk of developing symptomatic knee osteoarthritis is 40% in men and 47% in women; and the risk can be increased to 60% when the patient's BMI reaches 30 kg/m2. In this population, knee replacement is the most common, effective, and cost-effective method in all treatments with reducing pain, improving joint function and quality of life. Postoperative cognitive dysfunction (POCD) is a common complication in the elderly, and its incidence can reach 25-40% in major non-cardiac surgery. As for POCD can prolong hospital stay, increase mortality and morbidity, and increase social and economic burden, it is especially important for the prevention and treatment of POCD. However, The mechanism of POCD is still unclear. Studies suggest that it may involve inflammation and oxidative stress in the central nervous system. But for the elderly, they are in a state of low inflammatory response. At the same time, surgery and tourniquets also can trigger or aggravate inflammatory response. Once the inflammatory factors released into the blood circulation, they can act on the central nervous system in a variety of ways. As a result,elderly patients are more likely to develop POCD. In addition, some studies have shown that pain can also increase cognitive burden. Aspirin, its pharmacodynamic effects includes anti-inflammatory and analgesic effects which may have a certain effect on the prevention of POCD.

DETAILED DESCRIPTION:
Elderly patients undergoing knee replacement are more likely to develop POCD. The aim of this study is to determine the incidence of short-term POCD and long-term cognitive status in the elderly patients who use Aspirin atleast three months before knee replacement.And then, the study evaluates the effect of Aspirin on the incidence of postoperative delirium. In addition, it also shows the risk factors for POCD such as postoperative delirium, pain, C reactive protein and so on in the elderly patients who undergo knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 60 years old undergoing elective knee replacement with general anesthesia
* ASA score grade I-III
* Sign that informed consent is willing to participate in the study
* Can communicate in verbal
* The time of using aspirin is at least 3 months

Exclusion Criteria:

* Central nervous system disease;
* Mental illness before or now;
* With using Antipsychotic treatment such as sedatives or antidepressants;
* With drug dependence;
* Severe visual, auditory, or motor impairment;
* Acute infection;
* Emergency surgery;
* Serious systemic diseases;
* Preoperative delirium and/ or cognitive dysfunction preoperative;
* History of hospitalization 3 months before surgery.
* Participating in other research

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have major hemorrhoea perioperative, admitted to ICU postoperative and refuse participating the following up are screened out from the research.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of short-term POCD (Postoperative Cognitive Dysfunction) | within one week after surgery
  As measured by Mini-Mental State Examination

SECONDARY OUTCOMES:
Aspirin can increase the long-term cognitive function scores after surgery | at 1th month after surgery
  followed up by the Telephone Interview for Cognitive Status-Modified
The incidence of postoperative delirium | within one week after surgery
  As measured by the Confusion Assessment Method

CONTACTS AND LOCATIONS:
Overall Officials: Jindong Liu, M.S, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Murphy L, Schwartz TA, Helmick CG, Renner JB, Tudor G, Koch G, Dragomir A, Kalsbeek WD, Luta G, Jordan JM. Lifetime risk of symptomatic knee osteoarthritis. Arthritis Rheum. 2008 Sep 15;59(9):1207-13. doi: 10.1002/art.24021. PMID 18759314
- [Background] Price AJ, Alvand A, Troelsen A, Katz JN, Hooper G, Gray A, Carr A, Beard D. Knee replacement. Lancet. 2018 Nov 3;392(10158):1672-1682. doi: 10.1016/S0140-6736(18)32344-4. PMID 30496082
- [Background] Hasanain MS, Apostu D, Alrefaee A, Tarabichi S. Comparing the Effect of Tourniquet vs Tourniquet-Less in Simultaneous Bilateral Total Knee Arthroplasties. J Arthroplasty. 2018 Jul;33(7):2119-2124. doi: 10.1016/j.arth.2018.02.013. Epub 2018 Feb 15. PMID 29510953
- [Background] Ottens TH, Dieleman JM, Sauer AM, Peelen LM, Nierich AP, de Groot WJ, Nathoe HM, Buijsrogge MP, Kalkman CJ, van Dijk D; DExamethasone for Cardiac Surgery (DECS) Study Group. Effects of dexamethasone on cognitive decline after cardiac surgery: a randomized clinical trial. Anesthesiology. 2014 Sep;121(3):492-500. doi: 10.1097/ALN.0000000000000336. PMID 25225745
- [Background] Valentin LS, Pereira VF, Pietrobon RS, Schmidt AP, Oses JP, Portela LV, Souza DO, Vissoci JR, Luz VF, Trintoni LM, Nielsen KC, Carmona MJ. Effects of Single Low Dose of Dexamethasone before Noncardiac and Nonneurologic Surgery and General Anesthesia on Postoperative Cognitive Dysfunction-A Phase III Double Blind, Randomized Clinical Trial. PLoS One. 2016 May 6;11(5):e0152308. doi: 10.1371/journal.pone.0152308. eCollection 2016. PMID 27152422
- [Background] Steinmetz J, Christensen KB, Lund T, Lohse N, Rasmussen LS; ISPOCD Group. Long-term consequences of postoperative cognitive dysfunction. Anesthesiology. 2009 Mar;110(3):548-55. doi: 10.1097/ALN.0b013e318195b569. PMID 19225398
- [Background] Roach GW, Kanchuger M, Mangano CM, Newman M, Nussmeier N, Wolman R, Aggarwal A, Marschall K, Graham SH, Ley C. Adverse cerebral outcomes after coronary bypass surgery. Multicenter Study of Perioperative Ischemia Research Group and the Ischemia Research and Education Foundation Investigators. N Engl J Med. 1996 Dec 19;335(25):1857-63. doi: 10.1056/NEJM199612193352501. PMID 8948560
- [Background] Skvarc DR, Berk M, Byrne LK, Dean OM, Dodd S, Lewis M, Marriott A, Moore EM, Morris G, Page RS, Gray L. Post-Operative Cognitive Dysfunction: An exploration of the inflammatory hypothesis and novel therapies. Neurosci Biobehav Rev. 2018 Jan;84:116-133. doi: 10.1016/j.neubiorev.2017.11.011. Epub 2017 Nov 26. PMID 29180259